CLINICAL TRIAL: NCT06786507
Title: A Direct Head-to-head Comparison of Ustekinumab with Infliximab for the Treatment of Ulcerative Colitis
Status: Not yet recruiting | Type: Observational
Sponsor: Helwan University (Other)
Responsible Party: Principal Investigator, Myrna Mamdouh Sedki, Teaching assistant at Pharmacy Practice Department Faculty of Pharmacy - Helwan University, Helwan University
Other Study IDs: ustekinumab with infliximab
Record Dates: First submitted 2025-01-09; First posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Ulcerative Colitis (UC)
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Ustekinumab; Infliximab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- arm A is infliximab: for induction patients in this group will receive infliximab in week 0,2,6 for maintenance they will receive the drug every 8 weeks dose for both induction and maintenance is 5mg/kg IV
  Interventions: Drug: Infliximab
- arm B is ustekinomab: for induction patients in this group will receive an IV infusion with a weight based dose for maintenance they will receive a SC injection with a fixed dose 90mg every 8 weeks
  Interventions: Drug: Ustekinumab 90 mg

INTERVENTIONS:
Drug: Ustekinumab 90 mg — Ustekinumab is a human monoclonal IgG1 antibody that blocks the p40 subunit of both IL-12 and IL-23 this antagonistic action inhibits the interaction of these cytokines with the IL-12Rβ1 receptor. The IL-12Rβ1 receptor is found on the surface of NK cells and T cells which reduces inflammation and alters the body's immune response
  Groups: arm B is ustekinomab
Drug: Infliximab — Infliximab is a biological therapy/immunotherapy medication designed to stimulate the body's immune system and treat certain diseases. Infliximab is a purified, recombinant DNA-derived chimeric IgG monoclonal antibody protein that contains both murine and human components that inhibit tumor necrosis factor-alpha (TNF-α). TNF-α is a signaling protein involved in acute phase reactions and systemic inflammation. Macrophages, CD4+ lymphocytes, NK cells, neutrophils, mast cells, eosinophils, and neurons produce TNF-α. This TNF-α inhibition inhibits the inflammatory reaction's cascade, leading to improved disease condition inflammatory bowel disease
  Groups: arm A is infliximab

SUMMARY:
the goal of this study is to compare the efficacy of ustekinumab with infliximab for the treatment of ulcerative colitis aim of the study :

1. Compare effectiveness of ustekinumab versus infliximab therapy in remission achievement in UC patients.
2. Compare safety of ustekinumab therapy versus infliximab therapy in UC
3. To asses quality of life of ustekinumab therapy versus infliximab therapy in UC patients.

DETAILED DESCRIPTION:
Inflammatory bowel disease (IBD), including Crohn's disease (CD) and ulcerative colitis (UC), is a chronic inflammatory relapsing disorder affecting the gastrointestinal tract and is characterized by a progressive and unpredictable disease course.. The major subtypes are :

1. Crohn's Disease which affects any part of GIT.
2. Ulcerative Colitis which affects mainly the colon . And a subtype of IBD is called intermediate colitis (IC) when its unable to diffrentiate between UC and Crohns disease . There has been a global rise in the incidence of IBD over the last few decades, in 2017; there were 6.8 million cases of IBD globally. The age-standardized prevalence rate increased from 79.5 per 100, 000 population in 1990 to 84.3 per 100, 000 population in 2017. The annual incidence of Crohn's disease is 5.0 per 100,000 person-years in Asia and the Middle East, whereas incidence rates of ulcerative colitis are 6.3 per 100,000 person-years in Asia and the Middle East . some studies suggest the relative incidence ratio of UC and CD is 6:1 .Regarding UC the highest incidence of the disease is in Northern Europe and Canada at 24.3 and 19.2/100,000, respectively. Prevalence rates are also the highest in these two regions, at 505/100,000 in Northern Europe and 248/100,000 in Canada with incidence rate of 2.33 per 100,000 persons per year for UC in the Arab world Ulcerative colitis (UC) is a chronic, idiopathic inflammatory condition that affects the mucosa of the colon and rectum. Ulcerative colitis is also considered a progressive disease as it is associated with increased risk of disease extension, dysplasia/neoplasia, fibrosis and rectal dysfunction. Observational studies suggest that one-third of patients with left-sided colitis or disease limited to the rectum will develop pancolitis over a period of 10 years .

The changing epidemiology and the progressive nature of the disease require a clear understanding of the available and soon to become available therapeutic agents to treat UC and the different aspects of their pharmacology .

Treatments for inducing remission include 5-aminosalicylic acid drugs and corticosteroids. Maintenance treatments include 5-aminosalicylic acid drugs, thiopurines, biologics (eg,anti TNF , anti-cytokines and anti-integrins), and small molecules (Janus kinase inhibitors and sphingosine-1-phosphate receptor modulators) .

Infliximab is a biological therapy/immunotherapy medication designed to stimulate the body's immune system and treat certain diseases. Infliximab is a purified, recombinant DNA-derived chimeric IgG monoclonal antibody protein that contains both murine and human components that inhibit tumor necrosis factor-alpha (TNF-α). TNF-α is a signaling protein involved in acute phase reactions and systemic inflammation. Macrophages, CD4+ lymphocytes, NK cells, neutrophils, mast cells, eosinophils, and neurons produce TNF-α. This TNF-α inhibition inhibits the inflammatory reaction's cascade, leading to improved disease condition inflammatory bowel disease .

Infliximab has a high affinity for TNF-α and does not inhibit TNF-β. TNF-α is responsible for several physiological responses, including inducing proinflammatory cytokines (eg, IL-1 and IL-6), increasing adhesion molecule release, and enhancing the migration of leukocytes from blood vessels in the surrounding tissue (via increased endothelial permeability) . Infliximab is administered in dose 5 mg/kg i.v. for the whole induction and maintenance phase .

Ustekinumab is a human monoclonal IgG1 antibody that blocks the p40 subunit of both IL-12 and IL-23 this antagonistic action inhibits the interaction of these cytokines with the IL-12Rβ1 receptor. The IL-12Rβ1 receptor is found on the surface of NK cells and T cells which reduces inflammation and alters the body's immune response . ulcerative colitis treatment is based on an initial intravenous weight-based infusion followed by a subcutaneous maintenance schedule (90 mg subcutaneously eight weeks after initial intravenous administration and every eight weeks after that) .

The prognosis in UC is difficult to assess, however it should be emphasized that even one-third of patients need to undergo surgical treatment (colectomy) at different stages of the disease. Due to these data, together with the fact of increasing prevalence of UC reported in many industrialized and developing countries .

several treatment options now are available for the management of moderate-severe ulcerative colitis, with variable efficacy and safety profiles, and positioning different agents in the treatment course as first-line (in biologic-naïve patients) and second-line (in patients with prior exposure to tumor necrosis factor [TNF]-α antagonists) is a key knowledge gap. In the absence of head-to-head comparisons, prior network meta-analyses have attempted to address this gap, but have been limited by the number of studies especially at Egyptian population , that why this study will be conducted .

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are voluntarily able to give informed consent
* Subjects who can participate in all aspects of this clinical study
* Males and females aged from ≥ 18 to ≤ 80 years, at screening visit
* Diagnosis of moderate to severe UC established by clinical and endoscopic evidence.
* Biological therapy naïve patients.

Exclusion Criteria:

* - Previous exposure to IFX or UST or any other in IFX or UST-containing product
* Has a history of hypersensitivity or allergies to the ingredients of IFX or UST formulations
* Unstable angina
* Moderate or severe heart failure (defined as New York Heart Association Class III or IV)
* Chronic respiratory failure
* History of any major neurological disorders including stroke, multiple sclerosis, brain tumor, or neurodegenerative disease
* Chronic hepatitis B or C infection. Patients with positive viral serology at screening for infection with hepatitis B (HBV) or hepatitis C virus (HCV) may be eligible if the polymerase chain reaction test is negative, and the patients receive standard of-care antiviral prophylaxis (if applicable)
* Known severe chronic kidney failure
* Known severe chronic liver failure
* Known active or latent tuberculosis
* Ongoing HIV infection

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: moderate to severe ulcerative colitis bio naïve patients
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-05-15 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
(CRP) and Improvement degree of ulcerative colitis | baseline and after 6 months
  Efficacy that will be evaluated by:
  Degree of reduction in the level of inflammatory markers (CRP), Improvement degree of ulcerative colitis ( ≤5 mg/l)
safety evaluation | baseline and after 6 months
  Any adverse event will be reported by the patient for safety evaluation of both drugs will be analyzed.

SECONDARY OUTCOMES:
improvement in quality of life | baseline and after 6 months
  improvement in quality of life using IBDQ 32
  Secondary outcome definitions :The scores of patients range from 170 to 190.

CONTACTS AND LOCATIONS:
Locations (1):
- El-Demerdash hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: McDowell C, Farooq U, Haseeb M. Inflammatory Bowel Disease. [Updated 2022 Jun 27]. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2023 Jan. — https://pubmed.ncbi.nlm.nih.gov/29262182/
- See also: Alatab, S., Sepanlou, S. G., Ikuta, K., Vahedi, H., Bisignano, C., Safiri, S. ... & Alipour, V. (2020). The global, regional, and national burden of inflammatory bowel disease in 195 countries and territories, 1990-2017: a systematic analysis for the — https://pubmed.ncbi.nlm.nih.gov/31648971/
- See also: Elbadry M, Nour MO, Hussien M, Ghoneem EA, Medhat MA, Shehab H, Galal S, Eltabbakh M, El-Raey F, Negm M, Afify S, Abdelhamed W, Sherief A, Abdelaziz A, Abo Elkasem M, Mahrous A, Kamal G, Maher M, Abdel-Hameed O, Elbasuny A, El-Zayyadi I, Bassiony A, — https://pubmed.ncbi.nlm.nih.gov/35514748/
- See also: Mosli, M., Alawadhi, S., Hasan, F., Abou Rached, A., Sanai, F., & Danese, S. (2021). Incidence, Prevalence, and Clinical Epidemiology of Inflammatory Bowel Disease in the Arab World: A Systematic Review and Meta-Analysis. Inflammatory intestinal dise — https://pubmed.ncbi.nlm.nih.gov/34722642/
- See also: Le Berre, C., Honap, S., & Peyrin-Biroulet, L. (2023). Ulcerative colitis. Lancet (London, England), 402(10401), 571-584. — https://pubmed.ncbi.nlm.nih.gov/37573077/
- See also: Singh, S. Murad,M , Fumery M , Dulai ,P.S . Sandborn W .J.First- and Second-Line Pharmacotherapies for Patients With Moderate to Severely Active Ulcerative Colitis: An Updated Network Meta-Analysis Clinical Gastroenterology and Hepatology, Volume 18, — https://pubmed.ncbi.nlm.nih.gov/31945470/
- See also: Akiho H, Yokoyama A, Abe S, Nakazono Y, Murakami M, Otsuka Y, Fukawa K, Esaki M, Niina Y, Ogino H. Promising biological therapies for ulcerative colitis: A review of the literature. World J Gastrointest Pathophysiol. 2015 Nov 15;6(4):219-27. — https://pmc.ncbi.nlm.nih.gov/articles/PMC4644886/
- See also: You Y, Stelzl P, Joseph DN, Aldo PB, Maxwell AJ, Dekel N, Liao A, Whirledge S, Mor G. TNF-α Regulated Endometrial Stroma Secretome Promotes Trophoblast Invasion. Front Immunol. 2021;12:737401. — https://pubmed.ncbi.nlm.nih.gov/34790194/
- See also: Benson JM, Peritt D, Scallon BJ, Heavner GA, Shealy DJ, Giles-Komar JM, Mascelli MA. Discovery and mechanism of ustekinumab: a human monoclonal antibody targeting interleukin-12 and interleukin-23 for treatment of immune-mediated disorders. MAbs. 201 — https://pubmed.ncbi.nlm.nih.gov/22123062/
- See also: Sands BE, Sandborn WJ, Panaccione R, O'Brien CD, Zhang H, Johanns J, Adedokun OJ, Li K, Peyrin-Biroulet L, Van Assche G, Danese S, Targan S, Abreu MT, Hisamatsu T, Szapary P, Marano C., UNIFI Study Group. Ustekinumab as Induction and Maintenance The — https://pubmed.ncbi.nlm.nih.gov/31553833/